CLINICAL TRIAL: NCT01801813
Title: Observational Study of Risk Factors of Neuro-critical Care Complications Regarding Patients Undergoing Brain Tumour Neuro-surgery : a Prospective Validation of the Cranioscore.
Brief Title: Risk Factors of Complications Regarding Patients Undergoing Brain Tumour Neuro-surgery (Cranioscore).
Acronym: Cranioscore
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0416
Record Dates: First submitted 2013-02-15; First posted 2013-03-01 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2016-03

CONDITIONS: Neuro-surgery; Brain Tumor; Post-operative Complications; Neuro-ICU Stay
Keywords: Neuro-surgery; Post-operative complications; Neuro-ICU resources
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neurosurgery for brain tumor patients: Collecting pre-operative and per-operative data, neuro-radiological data and post-operative complications
  Interventions: Other: Collecting pre-operative, per-operative data, neuro-radiological data and post-operative neuro-surgery complications

INTERVENTIONS:
Other: Collecting pre-operative, per-operative data, neuro-radiological data and post-operative neuro-surgery complications

SUMMARY:
Patients undergoing a brain tumour neurosurgery with craniotomy may present rare but lifethreatening post-operative complications. There are currently no strong recommendations to help the clinician in an attempt to properly hospitalise these patients after their intervention (Neuro-ICU, ICU,surgical ward).

Determining risk factors of post-operative complications could optimise resources. Therefore hospitalisation in Neuro-ICU would be mandatory in only a little number of patients.

DETAILED DESCRIPTION:
Retrospective analysis of a prospective database to create a Risk Score. Post-operative neurosurgery complications recording (Hyponatremia < 135mmol/l,Insulin administration, Nausea-Vomiting, Glasgow Coma Score, Inhalation, Post-operative intra-cranial bleeding requiring neurosurgery, Intra-cranial hypertension, Use of osmotherapy, Status epilepticus, Brain death, Death).

Collection of datas as Duration of mechanical ventilation, Length of ICU stay, Length of hospital stay.

Validation of this score on an independent prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing neuro-surgery for a brain tumor

Exclusion Criteria:

* Neuro-surgical emergency

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing neuro-surgery for a brain tumor
Sampling Method: Non-Probability Sample
Enrollment: 795 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Post-operative complications requiring Neuro-ICU stay ≥ 24 hours after surgery for neurosurgical reason. | During ICU stay, average of 24 hours

SECONDARY OUTCOMES:
Describing post-operative complications in patients undergoing neuro-surgery for brain tumor. | During ICU stay, average of 24 hours
  Hyponatremia < 135mmol/l,Insulin administration, Nausea-Vomiting, Glasgow Coma Score, Inhalation, Post-operative intra-cranial bleeding requiring neurosurgery Intra-cranial hypertension, Use of osmotherapy, Status epilepticus, Brain death Death.
Duration of mechanical ventilation | Duration of mechinal ventilation, average of 12 hours
Length of ICU stay | Duration of ICU stay, average of 24 hours
Length of hospital stay | Duration of hospital stay, expected average 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Karim ASEHNOUNE, PhD, MD, Study Chair — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Background] Ziai WC, Varelas PN, Zeger SL, Mirski MA, Ulatowski JA. Neurologic intensive care resource use after brain tumor surgery: an analysis of indications and alternative strategies. Crit Care Med. 2003 Dec;31(12):2782-7. doi: 10.1097/01.CCM.0000098860.52812.24. PMID 14668615